CLINICAL TRIAL: NCT06618859
Title: Time-restricted Eating in Patients With Moderate Chronic Kidney Disease and Albuminuria: A Pilot Randomized, Open-label, Double-arm Trial (TRECK)
Brief Title: Time-restricted Eating in Patients With Moderate Chronic Kidney Disease and Albuminuria
Acronym: TRECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: de Seigneux Sophie (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, de Seigneux Sophie, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02172
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental)
  Interventions: Behavioral: Time-restricted eating
- Active control (Active Comparator)
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Time-restricted eating — Participants will be advised to consume meals and calorie-containing drinks only during a window of 8 hours, to be self-selected by the participant and advised by the investigators based on their daily routine and eating habits during the run-in phase.
  Other Names: TRE
  Arms: Time-restricted eating
Behavioral: Active control — Participants will be advised to keep the same eating rhythm and timing of meals per day during the intervention.
  Arms: Active control

SUMMARY:
Chronic kidney disease (CKD) affects approximately 12 to 15% of adults worldwide, with an increasing incidence expected. Major causes include diabetic nephropathy, hypertension, and various glomerulonephritis. Proteinuria is a key factor in identifying and assessing the risk of CKD progression.

The precise pathophysiology of CKD is not fully understood, but recent research highlights metabolic alterations, particularly in lipid and glucose metabolism. CKD progression is influenced by diet, as evidenced by recent studies. Interventions such as the ketogenic diet and time-restricted feeding show promising results in improving metabolism and may have beneficial effects on CKD.

Our study aims to evaluate the impact of time-restricted eating (TRE) on proteinuria, the decline in glomerular filtration rate, and weight loss in patients with moderate CKD with albuminuria (KDIGO stage 2-3). This will allow us to better understand the efficacy of this dietary approach tailored to the individual habits of participants.

The primary outcome measure will be albuminuria before and after the 12-week intervention. Secondary outcome measures will include the impact of fasting on blood pressure as assessed by 24-hour ambulatory monitoring, body composition evaluated by DXA and BIA, continuous glucose monitoring, and blood hormone profiles. Additionally, the feasibility and safety of TRE in this population will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria

  * Adult men and women
  * Chronic Kidney Disease with KDIGO stage G2 and G3 defined by a Glomerular Filtration Rate between 30 and 90 mL/min/1.73m2
  * Albuminuria stage A2 or A3, but without nephrotic-range proteinuria: 3 to 200 mg/mmol
  * Body mass index 18-40 kg/m2
  * Eating window of 12 hours (self-reported and measured during the run-in phase)
* Study-related criteria

  * Able to give informed consent and follow the study procedures for the entire duration
  * Confident use of a smartphone compatible with the MyFoodRepo app (iOS, Android) and able to take regular pictures of food/drinks

Exclusion Criteria:

* Clinical criteria

  * Pregnant and breastfeeding women, plans for maternity during the study
  * Eating disorder(s)
  * Other diets: low-carb, ketogenic diet, hypocaloric diets (eviction for food intolerances, vegan/vegetarian diet are not excluded)
  * Uncontrolled blood pressure (> 160/100 mmHg)
  * Diabetes with hypoglycemic drug(s) will be excluded, however those with impaired glucose tolerance (prediabetes, as defined by the American Diabetes Association) or diabetes with no risk of hypoglycemia (i.e. treated with non-hypoglycemic drugs or without medication) will be included
  * Oral corticosteroids
  * Uncontrolled diabetes HbA1c > 8.5%
  * Active cancer and/or oncologic treatment over the previous 12 months
  * Major mental illness
  * Consumption of > 7 standard units of alcohol per week for women and > 14 standard units of alcohol per week for men
  * Shift work, such as evening shifts or night shifts planned during the study
  * Travel/trip to a different time zone (≥ 2-hour time difference) planned during the study
* Study-related criteria and other interventions

  * Recent treatment modification in the last 3 months, including but not limited to ACE blockers, SLGT2i, finerenone
  * Patients with recent glomerulonephritis diagnosis on more than 2 immunosuppressive drugs
  * Patients with kidney transplant in the last past year
  * Enrolled in another interventional clinical trial (medication, medical device) over the previous 1 month and planned during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in urine albumin/creatinine ratio (UACR) | From randomization to close-out visit (12 weeks)
  Measured by 24h urine collection

SECONDARY OUTCOMES:
Change in creatinine- and cystatin-estimated glomerular filtration rate (eGFR) | From randomization to close-out visit (12 weeks)
  Measured in clinical chemistry
Change in blood pressure | From randomization to close-out visit (12 weeks)
  Measured by 24h ambulatory blood pressure monitoring (ABPM)
Change in systolic and diastolic blood pressure | From randomization to close-out visit (12 weeks)
  Measured with an arm cuff in the sitting position
Change in body fat mass and regional distribution | From randomization to close-out visit (12 weeks)
  Measured by dual-energy X-ray absorptiometry (DXA)
Change in body fat mass | From randomization to close-out visit (12 weeks)
  Measured by bioelectrical impedance (BIA)
Change in fasting glucose | From randomization to close-out visit (12 weeks)
  Measured in clinical chemistry
Change in glucose excursion | From randomization to close-out visit (12 weeks)
  Measured by continuous glucose monitoring (CGM)
Change in physical activity | From randomization to close-out visit (12 weeks)
  Measured by actigraphy
Change in sleep/wake cycles | From randomization to close-out visit (12 weeks)
  Measured by actigraphy
Change in sleep quality | From randomization to close-out visit (12 weeks)
  Measured by the Pittsburgh Sleep Quality Index (PSQI, range 0-21)
Change in eating duration | From randomization to close-out visit (12 weeks)
  Duration from the first to last caloric intake over the 24h cycle
Change in weight | From randomization to close-out visit (12 weeks)
  Body weight (kg)
Change in lipid profile (concentration of total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) | From randomization to close-out visit (12 weeks)
  Measured in clinical chemistry
Change in blood hormone profile | From randomization to close-out visit (12 weeks)
  Measured in clinical chemistry
Incidence of adverse events in response to the randomized intervention | From randomization to close-out visit (12 weeks)
  Adverse events graded after the Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sophie de Seigneux, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland